CLINICAL TRIAL: NCT01874080
Title: Bioequivalence Study of the Fixed Dosed Combination of 5 mg Saxagliptin and 1000 mg Metformin Extended Release Tablet Manufactured in Mt. Vernon, Indiana and Humacao, Puerto Rico Relative to the Fixed Dosed Combination Tablet Manufactured in Mt. Vernon, Indiana and Bioequivalence Study of the Fixed Dosed Combination of 5 mg Saxagliptin and 500 mg Metformin Extended Release Tablet Manufactured in Mt. Vernon, Indiana and Humacao, Puerto Rico Relative to the Fixed Dosed Combination Tablet Manufactured in Mt. Vernon, Indiana Administered to Healthy Subjects Under Fed Conditions
Brief Title: Bioequivalence Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CV181-208
Record Dates: First submitted 2013-06-06; First posted 2013-06-10 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-03

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — saxagliptin; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm A: Saxagliptin/Metformin XR FDC (Mt. Vernon/Humacao) (Experimental): Saxagliptin 5 mg /Metformin 1000 mg (Mt. Vernon/Humacao) tablet by mouth once daily on Day 1 of Periods 1 and 2
  Interventions: Drug: Saxagliptin/Metformin
- Arm B: Saxagliptin/Metformin XR FDC (Mt. Vernon) (Experimental): Saxagliptin 5 mg/Metformin 1000 mg (Mt. Vernon) tablet by mouth once daily on Day 1 of Periods 1 and 2
  Interventions: Drug: Saxagliptin/Metformin
- Arm C: Saxagliptin/Metformin XR FDC (Mt. Vernon/Humacao) (Experimental): Saxagliptin 5 mg/Metformin 500 mg (Mt. Vernon/Humacao) tablet by mouth once daily on Day1 of Periods 1 and 2
  Interventions: Drug: Saxagliptin/Metformin
- Arm D: Saxagliptin/Metformin XR FDC (Mt. Vernon) (Experimental): Saxagliptin 5 mg/Metformin 500 mg (Mt. Vernon) tablet by mouth once daily Day 1 of Periods 1 and 2
  Interventions: Drug: Saxagliptin/Metformin

INTERVENTIONS:
Drug: Saxagliptin/Metformin
  Other Names: Kombiglyze XR

SUMMARY:
The purpose of this study is to determine if tablets manufactured at different sites have the same bioavailability, that is yield similar blood levels/concentrations of the drugs and are handled by the body similarly

DETAILED DESCRIPTION:
Primary Purpose:

Other: Protocol designed to demonstrate the bioequivalence of the fixed dose combination of 5 mg Saxagliptin and 1000 mg Metformin Extended Release Tablet manufactured in Mt. Vernon, Indiana and Humacao, Puerto Rico relative to the fixed dose combination tablet manufactured in Mt. Vernon, Indiana and the bioequivalence of the fixed dose combination of 5 mg Saxagliptin and 500 mg Metformin Extended Release Tablet manufactured in Mt. Vernon, Indiana and Humacao, Puerto Rico relative to the fixed dose combination tablet manufactured in Mt. Vernon, Indiana in healthy human subjects under fed conditions

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects, 18-45 years of age
* Body mass index (BMI) of 18.0 to 30.0 kg/m2, inclusive
* Women must have a negative serum or urine pregnancy test within 24 hours prior to the start of investigational product

Exclusion Criteria:

* Any significant acute or chronic medical illness
* Estimated creatinine clearance of <60 mL/min as calculated using the Modification of Diet in Renal Disease method Current or recent (within 3 months of study drug administration)
* Gastrointestinal (GI) disease that could affect the absorption of study drug
* Inability to tolerate oral medication
* History of allergies or adverse reactions to DPP4 inhibitors or Metformin or related compounds
* Current smoker or recent (within 6 months of study drug administration) history of regular tobacco use (positive cotinine test)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2013-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Point estimates and 90% CIs for the ratio of geometric means for Cmax for Saxagliptin and Metformin in the 5/1000 mg FDC XR (Mt.Vernon/Humacao) and 5/1000 mg FDC XR (Mt. Vernon) | 19 time points up to Day 3 of Periods 1 and 2
  Cmax=Maximum observed plasma concentration
  CI=Confidence interval
  FDC=Fixed dosed combination
  XR=Extended release
Point estimates and 90% CIs for the ratio of geometric means for AUC(0-T) for Saxagliptin and Metformin in the 5/1000 mg FDC XR (Mt.Vernon/Humacao) and 5/1000 mg FDC XR (Mt. Vernon) | 19 time points up to Day 3 of Periods 1 and 2
  AUC(0-T)=Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration
Point estimates and 90% CIs for the ratio of geometric means for AUC(INF) for Saxagliptin and Metformin in the 5/1000 mg FDC XR (Mt.Vernon/Humacao) and 5/1000 mg FDC XR (Mt. Vernon) | 19 time points up to Day 3 of Periods 1 and 2
  AUC(INF)=Area under the plasma concentration-time curve from time zero extrapolated to infinity
Point estimates and 90% CIs for the ratio of geometric means for Cmax for Saxagliptin and Metformin in the 5/500 mg FDC XR (Mt. Vernon/Humacao) and 5/500 mg FDC XR (Mt. Vernon) | 19 time points up to Day 3 of Periods 1 and 2
Point estimates and 90% CIs for the ratio of geometric means for AUC(0-T) for Saxagliptin and Metformin in the 5/500 mg FDC XR (Mt. Vernon/Humacao) and 5/500 mg FDC XR (Mt. Vernon) | 19 time points up to Day 3 of Periods 1 and 2
Point estimates and 90% CIs for the ratio of geometric means for AUC(INF) for Saxagliptin and Metformin in the 5/500 mg FDC XR (Mt. Vernon/Humacao) and 5/500 mg FDC XR (Mt. Vernon) | 19 time points up to Day 3 of Periods 1 and 2

SECONDARY OUTCOMES:
Time to maximum observed plasma concentration (Tmax) for Saxagliptin and Metformin and for 5-OH Saxagliptin (Treatments A, B, C, and D) | 19 time points up to Day 3 of Periods 1 and 2
Terminal half life (T-HALF) for Saxagliptin and Metformin and for 5-OH Saxagliptin (Treatments A, B, C, and D) | 19 time points up to Day 3 of Periods 1 and 2
Cmax for 5-OH Saxagliptin (Treatments A, B, C, and D) | 19 time points up to Day 3 of Periods 1 and 2
AUC(0-T) for 5-OH Saxagliptin (Treatments A, B, C, and D) | 19 time points up to Day 3 of Periods 1 and 2
AUC(INF) for 5-OH Saxagliptin (Treatments A, B, C, and D) | 19 time points up to Day 3 of Periods 1 and 2
Safety assessments based on adverse event reports and the results of vital sign measurements, ECGs, physical examinations, and clinical laboratory tests | Up to Day 3 of Periods 1 and 2 and up to 30 days post discontinuation of dosing
  Parameters will include:
  1. Serious adverse events
  2. Deaths
  3. Adverse events leading to discontinuation
  4. Number of subjects with potentially clinically significant changes in vital signs, electrocardiograms (ECGs) or safety laboratory findings defined as meeting marked abnormality criteria

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Icon Development Solutions, San Antonio, Texas, United States

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: CV181208_CSR_Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3070&filename=CV181208_Synopsis.pdf